CLINICAL TRIAL: NCT03558048
Title: The Effect of Inflammatory Bowel Disease Flares on Serum Prostate Specific Antigen
Brief Title: The Effect of IBD Flares on Serum PSA
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: STU00207583
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases; Prostate Cancer
Keywords: Prostate Specific Antigen; IBD; PSA
MeSH Terms: conditions — Inflammatory Bowel Diseases; Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with Inflammatory Bowel Disease: Men with a confirmed diagnosis of IBD between the ages of 40-69 years old. These subjects will have their prostate specific antigen checked via a blood draw during clinic visits over the course of the study period.
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — Subjects will have their blood drawn during clinic visits over the course of the study period to measure their serum prostate specific antigen levels.

SUMMARY:
This study will measure Prostate Specific Antigen (PSA) values in men with Inflammatory Bowel Disease (IBD) before, during, and following a flare. In addition, the effect of any PSA increase will be analyzed and correlated to the location of disease (rectal vs. other). Study findings may help men with IBD by identifying pitfalls in prostate cancer screening for this population and help to stratify and understand the effect IBD has on the prostatic milieu. By optimizing how men with IBD are screened for prostate cancer, future unnecessary healthcare encounters and expenditures may be reduced for this patient group.

DETAILED DESCRIPTION:
Over one million adults in the U.S. are estimated to suffer from Inflammatory Bowel Disease (IBD), accounting for more than 2 million ambulatory and emergency room visits annually. This healthcare utilization may lead to an average increase of $5,000-$8,000 in annual medical expenditure per patient. Reducing unnecessary medical interactions and expenditures in this patient group is paramount and requires individualized disease monitoring and healthcare screening

One screening test that may lead to additional exams and costs is the Prostate Specific Antigen (PSA) test used to screen for prostate cancer. While PSA screening can reduce prostate cancer mortality, false-positive elevations are common, especially in the setting of non-malignant prostate inflammation. This research group recently reported in a large retrospective case-control series that after age 65, men with IBD who underwent prostate cancer screening at Northwestern Memorial Hospital (NMH) had higher serum PSA values than non-IBD controls. In addition, men with IBD had a significantly higher risk of clinically significant prostate cancer even when controlling for differences in PSA and other relevant covariates. However, whether the elevation in PSA is related to inflammation in these men with IBD versus a true reflection of an increased risk of prostate cancer is unclear. Furthermore, the interplay of IBD status and screening PSA values is currently unknown.

This study will measure PSA values in men with IBD before, during, and following a flare. In addition, the effect of any PSA increase will be analyzed and correlated to the location of disease (rectal vs. other). Study findings may help men with IBD by identifying pitfalls in prostate cancer screening for this population and help to stratify and understand the effect IBD has on the prostatic milieu. By optimizing how men with IBD are screened for prostate cancer, future unnecessary healthcare encounters and expenditures may be reduced for this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Men, ages 40-69 years old
* Confirmed diagnosis of IBD presenting to the Northwestern Memorial Hospital Gastroenterology Clinic

Exclusion Criteria:

* History of prostate cancer or prior prostate procedures (biopsies or transurethral resection)

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include men ages 40 to 69 presenting to the Northwestern Memorial Hospital Gastroenterology Clinic with a diagnosis of IBD. Men with a history of prostate cancer or prior prostate procedures (transurethral resection or biopsies) will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between IBD and PSA | 12 months
  Measure PSA values in men with IBD before, during, and following a flare

SECONDARY OUTCOMES:
Location of disease | 12 months
  Analyze and correlate PSA increase with location of disease

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans at this time to share individual participant data with other researchers. All patient identifying data will be removed prior to transfer to a statistician. No individual research subject will be identified in any reports from the study which will be statistical in nature.

REFERENCES:
- [Background] Kappelman MD, Moore KR, Allen JK, Cook SF. Recent trends in the prevalence of Crohn's disease and ulcerative colitis in a commercially insured US population. Dig Dis Sci. 2013 Feb;58(2):519-25. doi: 10.1007/s10620-012-2371-5. Epub 2012 Aug 29. PMID 22926499
- [Background] Ananthakrishnan AN, McGinley EL, Saeian K, Binion DG. Trends in ambulatory and emergency room visits for inflammatory bowel diseases in the United States: 1994-2005. Am J Gastroenterol. 2010 Feb;105(2):363-70. doi: 10.1038/ajg.2009.580. Epub 2009 Oct 6. PMID 19809414
- [Background] Kappelman MD, Rifas-Shiman SL, Porter CQ, Ollendorf DA, Sandler RS, Galanko JA, Finkelstein JA. Direct health care costs of Crohn's disease and ulcerative colitis in US children and adults. Gastroenterology. 2008 Dec;135(6):1907-13. doi: 10.1053/j.gastro.2008.09.012. Epub 2008 Sep 17. PMID 18854185
- [Background] Oesterling JE, Jacobsen SJ, Chute CG, Guess HA, Girman CJ, Panser LA, Lieber MM. Serum prostate-specific antigen in a community-based population of healthy men. Establishment of age-specific reference ranges. JAMA. 1993 Aug 18;270(7):860-4. PMID 7688054